CLINICAL TRIAL: NCT04146896
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of NYX-2925 in Subjects With Neuropathic Pain Associated With Diabetic Peripheral Neuropathy
Brief Title: Efficacy and Safety of NYX-2925 in Subjects With Neuropathic Pain Associated With Diabetic Peripheral Neuropathy (DPN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aptinyx (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NYX-2925-2008
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Results first posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Diabetic Peripheral Neuropathic Pain
MeSH Terms: interventions — NYX-2925

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive either placebo or NYX-2925.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization algorithm, randomization allocation, allocation to study drug or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NYX-2925 (Experimental): NYX-2925 50 mg
  Interventions: Drug: NYX-2925 50 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NYX-2925 50 mg — NYX-2925 administered orally
  Arms: NYX-2925
Drug: Placebo — Placebo administered orally
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of NYX-2925 versus placebo in treating the neuropathic pain associated with diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to assess the efficacy and safety of NYX-2925 in subjects with neuropathic pain associated with diabetic peripheral neuropathy.

The study will be a 13- to 16-week study, including a 1- to 4-week Screening Period, followed by a 12- week double-blind, randomized, placebo-controlled Treatment Period.

ELIGIBILITY:
Inclusion criteria:

* Informed consent
* Subject has diabetic peripheral neuropathy of symmetrical nature in lower extremities for ≥4 years and reports at least moderate pain over the last week
* Stable diabetic and protocol allowed medication during the study
* Agrees to use highly effective birth control during the study
* Has not participated in an interventional study for at least 30 days and agrees not to participate in another interventional study during the study

Exclusion Criteria:

* Pain due to other conditions or diseases that would complicate participation in the study or pain reporting
* Current or historical serious medical conditions
* Prior participation in NYX-2925 clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Aptinyx Clinical Site, Fresno, California
  - Aptinyx Clinical Site, Irvine, California
  - Aptinyx Clinical Site, Lomita, California
  - Aptinyx Clinical Site, Los Angeles, California
  - Aptinyx Clinical Site, Norco, California
  - Aptinyx Clinical Site, Pomona, California
  - Aptinyx Clinical Site, Santa Ana, California
  - Aptinyx Clinical Site, Tustin, California
  - Aptinyx Clinical Site, Brandon, Florida
  - Aptinyx Clinical Site, Clearwater, Florida
  - Aptinyx Clinical Site, Greenacres City, Florida
  - Aptinyx Clinical Site, Miami, Florida
  - Aptinyx Clinical Site, New Port Richey, Florida
  - Aptinyx Clinical Site, Tampa, Florida
  - Aptinyx Clinical Site, Winter Haven, Florida
  - Aptinyx Clinical Site, Winter Park, Florida
  - Aptinyx Clinical Site, Decatur, Georgia
  - Aptinyx Clinical Site, Marietta, Georgia
  - Aptinyx Clinical Site, Blackfoot, Idaho
  - Aptinyx Clinical Site, Flossmoor, Illinois
  - Aptinyx Clinical Site, Rochester, Michigan
  - Aptinyx Clinical Site, Hazelwood, Missouri
  - Aptinyx Clinical Site, Las Vegas, Nevada
  - Aptinyx Clinical Site, Brooklyn, New York
  - Aptinyx Clinical Site, New York, New York
  - Aptinyx Clinical Site, Rochester, New York
  - Aptinyx Clinical Site, Greenville, North Carolina
  - Aptinyx Clinical Site, Winston-Salem, North Carolina
  - Aptinyx Clinical Site, Duncansville, Pennsylvania
  - Aptinyx Clinical Site, Houston, Texas
  - Aptinyx Clinical Site, Mesquite, Texas
  - Aptinyx Clinical Site, Plano, Texas
  - Aptinyx Clinical Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NYX-2925: NYX-2925 50 mg QD
  NYX-2925 50 mg: NYX-2925 administered orally
- Placebo: Placebo QD
  Placebo: Placebo administered orally
Period: Overall Study
Arm/Group | NYX-2925 | Placebo
Started | 114 | 114
Completed | 97 | 92
Not Completed | 17 | 22
Not completed — Adverse Event | 5 | 8
Not completed — Lack of Efficacy | 3 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Non-compliance | 5 | 4
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Randomized in error | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NYX-2925 | Placebo | Total
Number analyzed (Participants) | 114 | 114 | 228
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (7.73) | 60.0 (8.63) | 60.8 (8.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 51 | 100
  Male | 65 | 63 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 47 | 89
  Not Hispanic or Latino | 72 | 67 | 139
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 27 | 48
  White | 86 | 80 | 166
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 114 | 114 | 228
Duration of DPN at Baseline (Years) [Mean (Standard Deviation); unit: years] | 8.593 (4.3059) | 8.701 (4.1238) | 8.647 (4.2065)

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Numeric Rating Scale (NRS) Score
Description: Change from baseline in the weekly mean of the daily Numeric Rating Scale (NRS) score assessing average pain intensity related to DPN in the past 24 hours. In the NRS, a participant selects a whole number (0 to 10) that best indicates the intensity of his/her pain, where 0 represents no pain and 10 represents worst pain imaginable.
Time Frame: Week 12
Population: Modified Intent to Treat Population includes all subjects who received at least one dose of study drug with at least one post-baseline assessment of the pain intensity NRS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NYX-2925 | Placebo
Number analyzed (Participants) | 113 | 112
units on a scale | -2.01 (1.821) | -2.27 (2.102)
Statistical Analysis 1: Comparison: NYX-2925 vs Placebo; Test type: Superiority; p = 0.704, t-test, 2 sided

2. Secondary Outcome: Daily Sleep Interference Scale (DSIS) Score
Description: Change from baseline in the weekly mean of the Daily Sleep Interference Scale (DSIS) scores. The DSIS asks participants to ''Select the number that best describes how much your pain has interfered with your sleep during the past 24 hours.'' Response options for the DSIS range from 0 (did not interfere with sleep) to 10 (completely interfered with sleep/unable to sleep due to pain).
Time Frame: Week 12
Population: Population Description: Modified Intent to Treat Population includes all subjects who received at least one dose of study drug with at least one post-baseline assessment of the pain intensity NRS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NYX-2925 | Placebo
Number analyzed (Participants) | 113 | 112
units on a scale | -2.11 (1.903) | -2.39 (2.344)
Statistical Analysis 1: Comparison: NYX-2925 vs Placebo; Test type: Superiority; p = .684, t-test, 2 sided

3. Secondary Outcome: Patient Global Impression of Change (PGI-C)
Description: Number of subjects 'much improved' or 'very much improved' on Patient Global Impression of Change (PGI-C)
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NYX-2925 | Placebo
Number analyzed (Participants) | 113 | 112
Participants | 38 | 40
Statistical Analysis 1: Comparison: NYX-2925 vs Placebo; Test type: Superiority; p = 0.743, t-test, 2 sided

4. Secondary Outcome: Number of Subjects Achieving ≥30% Pain Reduction
Description: Number of subjects achieving ≥30% pain reduction from baseline in the weekly mean NRS average pain intensity related to DPN
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NYX-2925 | Placebo
Number analyzed (Participants) | 113 | 112
Participants | 51 | 52
Statistical Analysis 1: Comparison: NYX-2925 vs Placebo; Test type: Superiority; p = .483, t-test, 2 sided

5. Secondary Outcome: Number of Subjects Achieving ≥50% Reduction
Description: Number of subjects achieving ≥50% reduction from baseline in the weekly mean NRS average pain intensity related to DPN
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NYX-2925 | Placebo
Number analyzed (Participants) | 113 | 112
Participants | 29 | 35
Statistical Analysis 1: Comparison: NYX-2925 vs Placebo; Test type: Superiority; p = .199, t-test, 2 sided

6. Secondary Outcome: Norfolk Quality of Life Questionnaire - Diabetic Neuropathy (QOL-DN) Score
Description: Change from baseline in the Norfolk Quality of Life Questionnaire - Diabetic Neuropathy (QOL-DN) score. The QOL-DN is a 47 item subject reported questionnaire. Scores range from 0-126, and lower scores indicate improved quality of life.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NYX-2925 | Placebo
Number analyzed (Participants) | 113 | 112
units on a scale | -15.3 (17.91) | -16.7 (21.14)
Statistical Analysis 1: Comparison: NYX-2925 vs Placebo; Test type: Superiority; p = .273, t-test, 2 sided

7. Secondary Outcome: Use of Rescue Medication
Description: Number of subjects using rescue medication
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NYX-2925 | Placebo
Number analyzed (Participants) | 113 | 112
Participants | 100 | 97
Statistical Analysis 1: Comparison: NYX-2925 vs Placebo; Test type: Superiority; p = .668, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events are defined as the start of the event occurring on or after the date of first dispensed study drug (Day 1, Baseline Visit) and before or on the last dose (Week 12). The protocol required adverse events to be followed to resolution of the adverse event.
Arm/Group | NYX-2925 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/114 | 2/114
Serious Adverse Events (participants affected / at risk) | 1/114 | 6/114
Other Adverse Events (participants affected / at risk) | 15/114 | 15/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NYX-2925 (N=114) | Placebo (N=114)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Non Cardiac Acute Chest Pain (General disorders) | 1 (1) | 0 (0)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Unstable Angina (Cardiac disorders) | 0 (0) | 1 (1)
Chronic kidney disease exacerbation (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Worsening of coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NYX-2925 (N=114) | Placebo (N=114)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 7 (7)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT04146896/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT04146896/SAP_001.pdf